CLINICAL TRIAL: NCT04979689
Title: Effects of Physical Rehabilitation With and Without Intensive Exercise Therapy of Shoulder External Rotators in Patients With Erb's Palsy
Brief Title: Intensive Therapy of Shoulder External Rotators in Erb's Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0204 Qurat
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Erbs Palsy
Keywords: external rotation, Intensive session, C5-C6
MeSH Terms: conditions — Brachial Plexus Neuropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive physical therapy (Experimental): Intensive session
  Interventions: Other: Intensive physical therapy
- Non intensive physical therapy (Other): Non intensive session
  Interventions: Other: Non intensive physical therapy

INTERVENTIONS:
Other: Intensive physical therapy — Intensive physical therapy treatment protocol was given for 3 months 3 times a week including 1.5- 2-hour session. Pre and post treatment assessments were taken. It included stretching for 20 min, Proprioception on ball for 20 minutes, quadruped for 10 min, vibration therapy for 20 min, tapping twice a month for 5 days, sensory therapy with beans for 20 min, supine lying with hand below head for 10-15 min, texturing for 15 min and activity of making tower with cups and hitting in outward direction for 15-20 min.
  Arms: Intensive physical therapy
Other: Non intensive physical therapy — Non intensive therapy included 45 min session 3 times a week for 3 months. Pre and post treatment assessments were taken. The protocol included stretching for 20 min, cross friction massage for 15 min, Ball catch and throw for 15 min. progression was made from light to heavy weight ball.
  Arms: Non intensive physical therapy

SUMMARY:
Erb's palsy is a common neurological injury occurs at the time of birth. It causes injury to the upper trunk nerve root c5-c6, i.e., supply is around shoulder and muscles of forearm and these nerves network from the spine and pass through the cervicoaxillary canal in the neck and the ribs and emerge into the axilla. Restoring external rotation in erb's palsy is quite difficult and mostly surgery is recommended but if physiotherapy sessions are given with extended time up to 2 hours and latest techniques are applied to strengthen external rotators then range of external rotation can be improved.

DETAILED DESCRIPTION:
Erb's palsy is form of brachial plexus palsy which involves injury to cervical nerve roots c5 c6 causing loss of movements and deformities i.e., internally rotated shoulder, hanging arm and waiter's tip hand deformity. Most common risk factors are shoulder dystocia, maternal obesity, breech presentation and high birth weight of child. Its incidence is 0.42 per 1000 live births in which 25% experience permanent impairment and injury.

Both Conservative and non-conservative treatment protocols are applied in erb's palsy but key interventions are positioning in early infancy, passive range of motions and gentle stretching. Another latest treatment approach is intensive physical therapy in which single session duration is extended to three to four hours with combination of treatments. This study will be randomized control trial, used to check effectiveness of intensive physical therapy to restore shoulder external rotation in erb's palsy. Subjects with erb's palsy meeting the predetermined inclusion and exclusion criteria will be divided into two groups by using lottery method. Pre assessment will be done by using AROM on goniometer as objective measurement. Subject in one group will be treated with intensive physical therapy and the other with conventional treatment. Each subject will receive 5 Treatment sessions per week for 6 months.

Recorded values will be analyzed by using SPSS version 25

ELIGIBILITY:
Inclusion Criteria:

* Children (male and female)
* Ages ranged from 9 months to 12 months
* Unilateral involvement of c5, c6 and c7
* patients did not undergo surgery of the nerves or plexus

Exclusion Criteria:

* Musculoskeletal or neuro-muscular abnormalities other than Erb's palsy
* Contractures or fixed limitations in the affected upper extremity
* Hypersensitivity to latex and adhesive tapes

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Modified MALLET scale | 12th weeks
  A scale of 1 to 5 is used to assess shoulder abduction, global external rotation, hand to neck, hand to back and hand to mouth position. An aggregate score is calculated by summing the 5 individual scores with a maximum score of 5.

SECONDARY OUTCOMES:
Goniometer | 12th Weeks, 5th day
  A goniometer is an instrument which measures the available range of motion at a joint.
  (Also mention all information which ROM u want to check) One BY one IN 4 and 5th number

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Ikram, MS, Principal Investigator — Riphah International University
Locations (1):
- Children Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] @article{basit2018erb, Palsy} T, author={Basit, Hajira and Ali, Citra Dewi M and Madhani NB, Year={2018}. Erbs Palsy
- [Background] Rahat S, Ahmad S, Bushra S. Role of physical therapy in improving the functional outcome of infants with Erb's palsy due to neurapraxia and Axonotmesis. Pakistan J Med Heal Sci. 2019;13(3):815-8.
- [Background] Afzal F, Afzal A. Effects of Conventional Combination Physical Therapy Treatment To Improve the Gross Motor and Functional Movements in Children With Erb'S Palsy. Int J Ther Rehabil Res. 2017;6(2):70.
- [Background] Sherief AAA. Electrical Stimulation Versus Arm Splint In Improving Fine More Skills In Erb's Palsy Children. Bull Fac Ph Th Cairo Univ. 2011;16(1):91-6.
- [Background] Said R, Ahmed S. KINESIO ARM TAPING AS PROPHYLAXIS AGAINST THE DEVELOPMENT OF ERB ' S ENGRAM Thesis Submitted in Partial Fulfillment of the Requirements for a Master Children and Its Surgery. 2004
- [Background] Malessy MJ, Pondaag W. Obstetric brachial plexus injuries. Neurosurg Clin N Am. 2009 Jan;20(1):1-14, v. doi: 10.1016/j.nec.2008.07.024. PMID 19064174
- [Background] Mazhar N, Hashmi M, Bashir S, Khan B, Khan S, Ahmad L. Physiotherapy & Physical Rehabilitation Prevalence of Erb ' s Palsy due to Shoulder Dystocia in Multan. 2019;4(3).
- [Background] Kc K, Shakya S, Zhang H. Gestational diabetes mellitus and macrosomia: a literature review. Ann Nutr Metab. 2015;66 Suppl 2:14-20. doi: 10.1159/000371628. Epub 2015 Jun 2. PMID 26045324
- [Background] Frade F, Gomez-Salgado J, Jacobsohn L, Florindo-Silva F. Rehabilitation of Neonatal Brachial Plexus Palsy: Integrative Literature Review. J Clin Med. 2019 Jul 5;8(7):980. doi: 10.3390/jcm8070980. PMID 31284431
- [Background] CK O. A Case of Erb-Duchenne Palsy in a Man, Aged 24. MOJ Anat Physiol. 2017;3(6):184-6.